CLINICAL TRIAL: NCT05500521
Title: Association Between Severe-to-profound Hearing Loss and the Vestibular Function of the Inner Ear
Brief Title: Association Between Severe-to-profound Hearing Loss and the Balance Function of the Inner Ear
Status: Enrolling by invitation | Type: Observational
Sponsor: Värmland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: Hearing-vestibular
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hearing Loss, Sensorineural, Severe; Hearing Loss, Sensorineural, Profound; Vestibular Disorder
Keywords: hearing loss; vestibular function; video head impulse test; VEMP; caloric irrigation; dizziness
MeSH Terms: conditions — Hearing Loss; Vestibular Diseases; Dizziness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe-to-profound hearing loss: Patients with severe-to-profound hearing loss will undergo investigation with caloric irrigation, video head impulse test and vestibular evoked myogenic potential. Patients will complete the Dizziness Handicap Inventory-questionnaire.
  Interventions: Diagnostic Test: Caloric irrigation; Diagnostic Test: vHIT; Diagnostic Test: VEMP
- Controls: Controls will undergo investigation with caloric irrigation, video head impuls test and vestibular evoked myogenic potential. Controls will complete the Dizziness Handicap Inventory-questionnaire.
  Interventions: Diagnostic Test: Caloric irrigation; Diagnostic Test: vHIT; Diagnostic Test: VEMP

INTERVENTIONS:
Diagnostic Test: Caloric irrigation — In a healthy ear irrigation with warm and cold water should give rise to an intense sensation of vertigo and involuntary eye movements called nystagmus. This nystagmus can be measured and thereby give an indication of the vestibular function in that ear.
Diagnostic Test: vHIT — This test measures the vestibular ocular reflex in all six semicircular canals (three in each ear). By performing a fast head thrust in the direction of the canal the eye response can be detected by a high-velocity video camera. A slower response indicates impaired function in that canal.
Diagnostic Test: VEMP — Utricular and saccular function can be measured by VEMP. Sound is presented in one ear at a time and the evoked myogenic potential in the sternocleidomastoid and the superior oblique muscles can be measured respectively. This gives a measurement of the function of the sacculus (cVEMP) and utriculus (oVEMP).

SUMMARY:
Severe-to-profound hearing loss can have a major impact on patients´ lives leading to social isolation and decreased quality of life. Most commonly the hearing loss is caused by damage to the inner ear or cochlear nerve. Since the vestibular system which is central for our balance is located in the inner ear it can be suspected that patients with severe-to-profound hearing loss also might have an impaired vestibular function. This impairment may lead to a feeling of dizziness or vertigo. This study aims to investigate if patients with severe-to-profound hearing loss also have impaired vestibular function. The vestibular function will be measured with caloric irrigation, video head impulse test and vestibular evoked myogenic potential.

DETAILED DESCRIPTION:
Background: It is well known that uncorrected hearing loss can lead to increased feeling of exhaustion, social isolation and decreased quality of life. Sensorineural hearing loss originates from a damage to the cochlea in the inner ear or to the cochlear nerve and progresses with increasing age. Severe-to-profound hearing loss (STPHL) is defined as hearing levels 70 dB or worse on the better ear. The Swedish registry for adult patients with STPHL has showed that 30 % of the patients suffer from vertigo or dizziness often or always. The reasons for this are not established.

Apart from the cochlea the inner ear harbors the vestibular system consisting of the semicircular canals and the two otolithic organs, utriculus and sacculus. The vestibular system is the sensory system that helps us maintain balance. This study aims to investigate if patients with STPHL ie cochlear injury also have impaired vestibular function ie damage to the vestibular system.

The function of the vestibular system can be measured in three main ways. The semicircular canals can be assessed with caloric irrigation and video head impulse test (vHIT). The function of the sacculus and utriculus can be determined by the recording of vestibular evoked myogenic potential (VEMP). The sacculus is assessed by cervical VEMP (cVEMP) and the utriculus by ocular VEMP (oVEMP).

In patients with sensorineural STPHL the damage is most often located in the cochlea in the inner ear. The hypothesis in this study is that these patients also have a deteriorated function in the vestibular system. The aim of this study is to investigate whether the vestibular function between persons with STPHL

Method: This study will be conducted in the county of Värmland in Sweden, a county with approximately 280,000 inhabitants. Auditbase is the hearing data software used in Värmland where all audiograms are stored. By conducting a database search The investigators have identified all patients in Värmland with severe-to-profound hearing loss.

Patients aged 50-85 years have been extracted from the initial pool of patients. Ethical approval has been gained from the Ethics Review Authority in Sweden. An invitation will be sent to these patients. Only patients with a strict sensorineural hearing loss will be included in the study. Patients with a cochlear implant will be excluded. After a signed informed consent has been retrieved from the patient a time for testing will be scheduled.

The patient will undergo testing with caloric irrigation, vHIT and VEMP. Prior to testing patient will undergo an otoscopy to verify an intact eardrum.

The tests are described in detail below.

Caloric irrigation: Bi thermal caloric irrigation is performed with 30 and 44 degree water. Eye movements are recorded with goggles that prevent visual fixation.Nystagmus is recorded for ten seconds prior to irrigation. Irrigation then follows for a total of 30 seconds. Nystagmus is then recorded during one minute followed by 10 seconds with fixation and finally 10 seconds without fixation. Slow phase velocity (SPV) is automatically calculated for each irrigation. Since both ears are measured with cold and warm water four SPV-values are recorded.

VHIT: This test is carried out in a well-lit room with the patient seated in a height-adjustable, rotatable chair. Fast head thrusts are performed in the direction of the semicircular canal. A high speed camera detects the head movement and the corresponding eye response is recorded. This gives a measurement of the vestibulo-ocular reflex in the tested canal. If the eye response matches the speed of the head movement the resulting gain value will be close to 1. With a slower eye response the gain value will decrease indicating impaired function in that canal.

VEMP: Utricular and saccular function can be measured by VEMP. Sound (500 Hz toneburst, 124 dB SPL) is presented in one ear at a time and the evoked myogenic potential in the sternocleidomastoid and the superior oblique muscles can be measured respectively. This gives a measurement of the function of the sacculus (cVEMP) and utriculus (oVEMP). The measurements that can be performed and analyzed are: response (yes/no), latency to the response and, amplitude of the response.

The results of the tests will be used to compare whether there are any detectable differences between patients with STPHL and the control group without STPHL.

ELIGIBILITY:
Inclusion Criteria:

* Hearing level of 70 decibel or worse in the better ear

Exclusion Criteria:

* Congenital deafness
* Presence of cochlear implant/implants
* Severe vision impairment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up by 50 patients with severe-to-profound hearing loss and 50 age-matched controls with age-adequate hearing levels.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Video head impuls test (vHIT) | Baseline
  The vHIT gives a gain value of the vestibulo-ocular reflex for each of the semicircular canals. The values of patients with STPHL will be compared with the values from the controls.
Cervical vestibular evoked myogenic potential (cVEMP). | Baseline
  cVEMP gives information whether the response can be recorded at all. The latency time to the response and the amplitude of the response will be measured. The values of patients with STPHL will be compared with the values from the controls.
Ocular vestibular evoked myogenic potential (oVEMP). | Baseline
  oVEMP gives information whether the response can be recorded at all. The latency time to the response and the amplitude of the response will be measured. The values of patients with STPHL will be compared with the values from the controls.
Caloric irrigation | Baseline
  This tests results in two measurements of slow phase velocity of the nystagmus in each ear. A total of four measurements when combining both ears. The values of patients with STPHL will be compared with the values from the controls.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Inge Carlsson, PhD, Principal Investigator — University of Örebro, Faculty of medicine and health
Locations (1):
- Department of otorhinolaryngology, Karlstad, Sweden